CLINICAL TRIAL: NCT00422071
Title: Detecting a Reward Signal in the Motor Cortex
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070063; 07-N-0063
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-03-06

CONDITIONS: Healthy
Keywords: Transcranial Magnetic Stimulation (TMS); Dopamine; Gambling; Healthy Volunteer; HV
MeSH Terms: conditions — Gambling

SUMMARY:
This study will use transcranial magnetic stimulation (TMS) to determine whether the activity in the brain when someone wins something affects the part of the brain that controls movement. Studies have shown that the brain releases signals to mark rewards for certain behavior, like the activity the brain generates when an animal receives food or drink after performing a certain action. This study will look for a way to detect this kind of signal in humans.

Healthy volunteers between 18 and 60 years of age are eligible for this study. Participants undergo TMS during two experiments slot machine stimulation and key sequence (see below). For TMS, a wire coil is held on the subject s scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The stimulation may cause twitching in muscles of the face, arm or leg, and there may be a pulling sensation on the skin under the coil. The effect of TMS on the muscles is detected with small metal disk electrodes taped onto the skin of the arms or legs.

The stimulation strength needed to activate the hand muscles is determined at the beginning of each experiment. To do this, the subject sits with his or her arms and hand relaxed. Magnetic pulses of varying strengths are applied in order to find the right strength. Also, a series of 45 pairs of magnetic pulses is administered so close to each other that they produce only one movement. Measurements of the movements generated serve as a baseline for comparison with movements generated during the experiments.

Slot Machine Simulation

Subjects play a computer game similar to a slot machine. They press a button to start the game and watch as three barrels of the machine spin into place. Subjects can win $0.25, $1or $5 if all three barrels match when they stop spinning. If all three barrels do not match, subjects do not win any money, except in rare instances, when they are awarded money even when all three barrels do not match. In one trial in this experiment, subjects receive transcranial magnetic stimulation after they see the second barrel stop spinning. In another trial, they receive the stimulation after the third barrel stops spinning.

Key Sequence

Subjects see a letter on a computer screen and press a combination of the three keyboard keys G, H, and J. If they press the keys in the right order and under the time limit, they win $1. At some point, the letter displayed changes, and the subjects must guess a new combination to earn money. Each of the letters corresponds to its own combination of key presses. A few moments after the subjects see whether they pressed the keys in the right order, they receive TMS.

DETAILED DESCRIPTION:
Objectvie:

The role of mesencephalic dopamine neurons in reward processing has been established in primates using electrophysiological techniques and in humans using functional neuroimaging. Their role is thought to be dual: i) they show sustained activity with the expectation of a future reward and ii) a phasic response after reward. Animal data indicate that these neurons, located in the midbrain areas A8-10, behave as a single functional unit when activated. They have rich projections to both the prefrontal and motor cortices where they synapse on interneurons and cortical pyramidal cells, producing primarily inhibition. Though their function is not fully understood, these projections clearly play an important role in motivation and learning. Since there are no electrophysiological techniques available to detect dopaminergic or inhibitory activity in the human prefrontal cortex, our objective is to develop a paradigm to detect a reward related signal in the primary motor cortex, where transcranial magnetic stimulation can be used to measure brief events.

Study Population:

The population that we will study will be healthy volunteers between the ages of 18-60, without any significant medical history, contraindication to TMS or history of addictive behavior.

Design:

Our hypothesis is that the dopamine reward-related signal will alter level of evocable inhibition in primary motor cortex. Using behavioral paradigms that deliver intermittent reward, we aim to demonstrate a difference in the amount of cortical inhibition, i) when reward is expected compared to when reward is not expected ii) after rewarded compared to unrewarded trials iii) when reward follows a variable effortful response, and iv) when there is uncertainty as to whether a reward will be administered. If we are unable to produce a signal in the motor cortex with these simple paradigms, we will look for a reward-related change in inhibition when the rewarded behavior is the associative learning of a motor sequence. We will control for effects of variations in attention related to the experimental task, but not specific for reward, with a similar behavioral paradigm that manipulates attention and expectation.

Outcome Measures:

The outcome measures will be changes in the conditioned/unconditioned MEP for each reward condition.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women, age 18-60.

EXCLUSION CRITERIA:

Significant neurological or psychiatric history.

History of habitual gambling, defined as either visiting casinos more than once per month or playing cards for money more than once per week or gambling over the internet more than once per month.

Habitual consumption of more than two drinks a day, marijuana more than once a week or any other illicit drug use within the last three months.

Use of medication affecting the DA system, such as phenothiazine antihistamines (promethazine), antiemetics or decongestants within the last month.

Seizure History.

Significant abnormality on neurological examination.

Metal in the cranial cavity or eye, pacemaker, implanted pumps or stimulators.

Subjects who have participated in experiments 1-5 in this protocol may not participate in experiment 6, or 7.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2007-01-08; Study Completion 2014-03-06

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Avanzi M, Uber E, Bonfa F. Pathological gambling in two patients on dopamine replacement therapy for Parkinson's disease. Neurol Sci. 2004 Jun;25(2):98-101. doi: 10.1007/s10072-004-0238-z. PMID 15221629
- [Background] Cohen MX, Young J, Baek JM, Kessler C, Ranganath C. Individual differences in extraversion and dopamine genetics predict neural reward responses. Brain Res Cogn Brain Res. 2005 Dec;25(3):851-61. doi: 10.1016/j.cogbrainres.2005.09.018. Epub 2005 Nov 11. PMID 16289773
- [Background] Strobel A, Spinath FM, Angleitner A, Riemann R, Lesch KP. Lack of association between polymorphisms of the dopamine D4 receptor gene and personality. Neuropsychobiology. 2003;47(1):52-6. doi: 10.1159/000068876. PMID 12606846